CLINICAL TRIAL: NCT01530698
Title: Single-step Antigen Loading and TLR Activation of Dendritic Cells by mRNA Electroporation for Vaccination in Stage III and IV Melanoma Patients
Brief Title: Single-step Antigen Loading and TLR Activation of Dendritic Cells in Melanoma Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL2009-015737-73; 2009-015737-73 (EudraCT Number); AMO2009-084 (Other: Radboud University Nijmegen Medical Centre)
Record Dates: First submitted 2011-03-31; First posted 2012-02-10 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2014-11

CONDITIONS: Melanoma
Keywords: dendritic cell vaccination; melanoma; toll like receptor ligands; mRNA electroporation; vaccines
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- single step DC treatment (Experimental): vaccination with autologous dendritic cells treated with mRNA electroporation for single-step antigen loading and TLR activation (TriMix-DC)
  Interventions: Biological: autologous dendritic cell vaccine
- two step DC treatment (Active Comparator): vaccination with autologous dendritic cells treated with mRNA electroporation for antigen loading and separately for TLR activation
  Interventions: Biological: autologous dendritic cell vaccine

INTERVENTIONS:
Biological: autologous dendritic cell vaccine — Autologous monocyte-derived dendritic cells electroporated with mRNA encoding gp100 and tyrosinase (for antigen loading), active TLR4 and CD70 (for activation). Dendritic cells are vaccinated intranodally 3 times with biweekly intervals every 6 months, if no signs of progression, for a total of 9 vaccinations
  Arms: single step DC treatment
Biological: autologous dendritic cell vaccine — Autologous monocyte-derived dendritic cells electroporated with mRNA encoding gp100 and tyrosinase and matured with either cytokines or TLR ligands. Dendritic cells are vaccinated intranodally 3 times with biweekly intervals every 6 months, if no signs of progression, for a total of 9 vaccinations
  Arms: two step DC treatment

SUMMARY:
Objectives: This is an exploratory study, consisting of two parts. In part I dose escalation is performed and the primary objective is the safety of different doses of TLR-DC and Trimix DC. In part II Trimix DC vaccination will be compared with TLR-DC vaccination and the primary objective of this part is the immunological response, with toxicity and clinical efficacy being secondary objectives. These studies will provide important data on the safety and immunological effects of TLR-DC and Trimix DC.

Study design: Part I of this study is an open label dose escalation study. Part II of this study is an open label randomized phase II study.

Study population: Our study population consists of melanoma patients, with proven expression of melanoma associated tumor antigens gp100 and tyrosinase. Melanoma patients with regional lymph node metastasis in whom a radical lymph node dissection is performed within 2 months of inclusion in this study (further referred to as stage III) and melanoma patients with measurable distant metastases (further referred to as stage IV) will be included.

DETAILED DESCRIPTION:
1. Rationale Immunotherapy applying ex vivo generated and tumor-antigen-loaded dendritic cells (DC) has now successfully been introduced in the clinic. A limited, but consistent, number of objective immunological and clinical responses have been observed. Thusfar it remains unclear why some patients respond and others not, but there is a general consensus that the current protocols applied to generate DC may not result in the induction of optimal Th1 responses. The investigators and others have demonstrated that DC maturation is one of the crucial factors, not only for effective DC migration but also to induce effective anti-tumor immune responses in cancer patients. Currently, the "golden standard" used to mature DC consists of a cocktail of pro-inflammatory cytokines (IL-1b, IL-6, TNFa) and prostaglandin E2 (PGE2). Recent mouse data demonstrated, however, that maturation of DC by solely pro-inflammatory cytokines yielded DC that supported T cell clonal expansion, but failed to efficiently direct effector T cell differentiation. Interestingly, DC matured in the presence of Toll like receptor (TLR) ligands were able to induce full T cell effector function and unleashed more potent immune responses. The investigators recently identified vaccines against infectious diseases that contain TLR ligands and are capable of inducing DC maturation. This knowledge provides a new application for these clinical applicable agents: clinical grade DC stimulators. A clinical grade DC maturation protocol is developed in which TLR ligands (preventive vaccines) and PGE2 are combined which resulted in the generation of mature DC that secrete high levels of the key cytokine IL-12. Moreover, these TLR-ligand matured DC (TLR-DC) induced T cells secreting at least 20-fold higher levels of the effector cytokines IFNa and TNFa as compared to DC matured in the absence of TLR ligands.

   In the group of Kris Thielemans and it was shown that the T-cell stimulatory capacity of peptide-pulsed DC can be greatly enhanced by providing them with three different molecular adjuvants through electroporation with mRNA encoding a so-called TriMix of CD40 ligand (CD40L), CD70, and a constitutively active form of TLR4 (caTLR4). The combination of CD40L and caTLR4 electroporation would mimic CD40 ligation and TLR4 signaling of the DC and generates phenotypically mature, cytokine/chemokine-secreting DC, as has been shown for CD40 and TLR4 ligation through addition of soluble CD40L and lipopolysaccharide. On the other hand, the introduction of CD70 into the DC would provide a costimulatory signal to CD27+ naive T cells by inhibiting activated T cell apoptosis and by supporting T cell proliferation.

   In conclusion, these in vitro data demonstrate that both TLR-DC and Trimix DC are promising candidates to improve immunological and clinical responses in cancer immunotherapy.
2. Objectives This is an exploratory study, consisting of two parts. In part I dose escalation is performed and the primary objective is the safety of different doses of TLR-DC and Trimix DC. In part II Trimix DC vaccination will be compared with TLR-DC vaccination and the primary objective of this part is the immunological response, with toxicity and clinical efficacy being secondary objectives. These studies will provide important data on the safety and immunological effects of TLR-DC and Trimix DC.
3. Study design Part I of this study is an open label dose escalation study. Part II of this study is an open label randomized phase II study.
4. Study population Our study population consists of melanoma patients, with proven expression of melanoma associated tumor antigens gp100 and tyrosinase. Melanoma patients with regional lymph node metastasis in whom a radical lymph node dissection is performed within 2 months of inclusion in this study (further referred to as stage III) and melanoma patients with measurable distant metastases (further referred to as stage IV) will be included.
5. Main study endpoints The primary objectives of the study are to investigate the toxicity of TLR-DC and Trimix DC by dose escalation of DC numbers in part I, and to investigate immunological responses upon DC vaccination in part II of the study.

Immunological responses are:

1. The activation of immune cells in vivo.
2. The immunological response induced with TLR-DC and Trimix DC loaded with mRNA encoding melanoma-associated tumor antigens (gp100 and tyrosinase).

Safety and clinical efficacy are secondary objectives.

ELIGIBILITY:
Inclusion Criteria:

(All patients):

* histologically documented evidence of melanoma
* stage III or IV melanoma according to the 2001 AJCC criteria
* melanoma expressing gp100 (compulsory) and tyrosinase (non-compulsory)
* WHO performance status 0-1 (Karnofsky 100-70)
* life expectancy ≥ 3 months
* age 18-70 years
* no clinical signs or symptoms of CNS metastases
* WBC > 3.0x10e9/l, lymphocytes > 0.8x10e9/l, platelets > 100x10e9/l, serum creatinine < 150 µmol/l, serum bilirubin < 25 µmol/l
* normal serum LDH (< 450 U/l)
* expected adequacy of follow-up
* no pregnant or lactating women
* written informed consent

(Stage III melanoma)

* radical regional lymphnode dissection is performed (Stage IV melanoma)
* at least one unidimensional measurable target lesions according to RECIST, not previously irradiated, and no significant symptoms of disease requiring other palliative treatments

Exclusion Criteria:

* prior chemotherapy, immunotherapy or radiotherapy < 4 weeks prior to planned vaccination or presence of treatment-related toxicity
* history of any second malignancy in the previous 5 years, with the exception of adequately treated basal cell carcinoma or carcinoma in situ of the cervix
* serious active infections, HbsAg or HIV positive or autoimmune diseases or organ allografts
* concomitant use of immunosuppressive drugs
* known allergy to shell fish (since it contains KLH)
* rapidly progressive symptomatic disease
* any serious clinical condition that may interfere with the safe administration of DC

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-04; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
The primary objective of the study isto investigate immunological responses upon vaccination | 3 years
  The immunological response induced with TLR-DC and Trimix DC loaded with mRNA encoding melanoma-associated tumor antigens (gp100 and tyrosinase) will be evaluated by using 1. tetramer screening of skin-test biopsy derived cell-cultures and peripheral blood, 2. cytokine-bead assay to measure specific cytokine production of skin-test biopsy derived cell-cultures upon differential stimulation and 3. KLH-specific antibody and proliferative responses
The second primary objective is the toxicity of TLR-DC and Trimix-DC | 3 years
  toxicity will be reported with regard to 1. flu-like symptoms, 2. local injection site reaction and 3. other signs and symptoms, graded according to CTC version 3.0, numbers of patients and CTC grade will be reported

SECONDARY OUTCOMES:
clinical efficacy | 5 years
  progression free survival

CONTACTS AND LOCATIONS:
Overall Officials: C.J.A. Punt, prof.dr., Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands

REFERENCES:
- See also: Radboud University Nijmegen Medical Centre, Dept of Medical Oncology — http://www.umcn.nl
- See also: Nijmeegs Offensief Tegen Kanker — http://www.notk.nl
- See also: Central Committee on Research involving Human Subjects (CCMO), The Netherlands — http://www.ccmo.nl